CLINICAL TRIAL: NCT02741128
Title: Safety and Immunogenicity of a Tetravalent Dengue Vaccine in HIV-Positive Adults Aged 18 to 50 Years in Brazil
Brief Title: Safety and Immunogenicity of a Tetravalent Dengue Vaccine in HIV-Positive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CYD50; U1111-1174-4398 (Other: WHO)
Record Dates: First submitted 2016-04-08; First posted 2016-04-18 (Estimated); Results first posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-01

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Human Immunodeficiency Virus
Keywords: Dengue Fever; Dengue Hemorrhagic Fever; Human Immunodeficiency Virus; CYD Dengue Vaccine
MeSH Terms: conditions — Dengue; Severe Dengue; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CYD Dengue vaccine group (Experimental): Subjects will receive 3 doses of CYD dengue vaccine at 0, 6, and 12 months
  Interventions: Biological: CYD Dengue Vaccine
- Placebo vaccine group (Placebo Comparator): Subjects will receive 3 doses of placebo (NaCl, 0.9%) vaccine at 0, 6, and 12 months
  Interventions: Biological: Placebo (NaCl 0.9%) vaccine group

INTERVENTIONS:
Biological: CYD Dengue Vaccine — 0.5 mL, Subcutaneous at Day 0, 6 and 12 months, respectively
  Arms: CYD Dengue vaccine group
Biological: Placebo (NaCl 0.9%) vaccine group — 0.5 mL, Subcutaneous at Day 0, 6 and 12 months, respectively
  Arms: Placebo vaccine group

SUMMARY:
The aim of the study was to evaluate the safety and immunogenicity of the Dengue vaccine in a population of special interest, such as HIV-positive adults previously exposed to dengue.

Primary Objective:

* To describe the safety of each injection of CYD dengue vaccine in HIV-positive adults previously exposed to dengue.

Secondary Objectives:

* To describe the humoral immune response to each dengue serotype at baseline and after each injection of CYD dengue vaccine in HIV-positive adults previously exposed to dengue.
* To detect the CYD dengue vaccinal viremia post-Inj 1 in HIV-positive adults previously exposed to dengue.
* To describe changes in CD4 count and HIV RNA viral load after each injection of CYD dengue vaccine in HIV-positive adults previously exposed to dengue.

Observational Objective:

* To describe the FV (YF, Dengue, Zika) serological status in the study population at baseline.

DETAILED DESCRIPTION:
Eligible subjects were randomized in a 2:1 ratio into 1 of 2 groups to receive 3 injections of either CYD dengue vaccine or placebo at 0, 6, and 12 months. The enrollment of subjects was carried out in two steps, including an early safety data review before the second step. The duration of each subject's participation in the study was approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 50 years on the day of first study vaccination (study product administration) ("18 to 50" means from the day of the 18th birthday to the day before the 51th birthday)
* Inform concent form has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* Documented seropositivity for HIV-1 infection based on the Brazilian HIV Guidelines' laboratory criteria (i.e., two positive results obtained from different and independent determination methods) or detectable HIV-1 viral load results in the past
* Stable HIV condition according to Brazilian HIV Guidelines (i.e., with both CD4 count > 350 cells/mm3 and sustainable and undetectable HIV viral load [< 50 copies/mL]) for at least 1 year before consent
* Stable antiretroviral (ART) regimen based on local HIV protocol for at least 1 year before consent.
* Previous exposure to dengue confirmed by rapid diagnostic test (RDT) or dengue IgG ELISA

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination)
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Previous vaccination against dengue disease with either the trial vaccine or another vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Self-reported or suspected congenital or acquired immunodeficiency, except HIV; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Previous acquired immunodeficiency syndrome (AIDS), defined as the occurrence of opportunistic infection in the last 2 years before consent
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the trial or to a vaccine containing any of the same substances
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Moderate or severe acute illness/infection (according to investigator judgment) or febrile illness (temperature ≥ 38.0°C) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Previous CD4 count < 200 cells/mm3 (nadir) since diagnosis of HIV
* History of chronic and active hepatitis B infection or HBsAg-positive
* History of chronic and active hepatitis C infection or HCV Ab-positive
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), urea and creatinine > 3 times the upper limit of normal range (ULN)
* Hemoglobin (Hb) < 10 g/dL
* White blood cell count (WBC) < 1500 cells/mm3
* Platelets < 100,000 cells/mm3.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (4):
- Brazil (4):
  - Investigational Site Number :0760002, Nova Iguaçu, Rio de Janeiro
  - Investigational Site Number :0760004, Natal, Rio Grande do Norte
  - Investigational Site Number :0760001, São Paulo
  - Investigational Site Number :0760003, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 centers in Brazil from 06 November 2019 to 07Jul 2021.
Pre-assignment Details: A total of 133 participants were randomized in 2:1 ratio of which 132 participants received vaccination.
Groups:
- CYD Dengue Vaccine: Participants were administered a single dose of subcutaneous (SC) injection of live, attenuated, tetravalent CYD dengue vaccine each on Day 0, 6 months and 12 months.
- Placebo: Participants were administered a single dose of SC injection of placebo vaccine each on Day 0, 6 months and 12 months.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine | Placebo
Started | 89 | 44
Vaccinated | 88 | 44
Completed | 82 | 43
Not Completed | 7 | 1
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety analysis set (SafAS) consisted of participants who had received study vaccine and for which safety data were scheduled to be collected.
Groups:
- CYD Dengue Vaccine: Participants were administered a single dose of SC injection of live, attenuated, tetravalent CYD dengue vaccine each on Day 0, 6 months and 12 months.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine | Placebo | Total
Number analyzed (Participants) | 88 | 44 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.8 (7.60) | 36.3 (7.88) | 36.7 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 20 | 51
  Male | 57 | 24 | 81
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Unsolicited Systemic Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant administered study vaccine and which did not necessarily have a causal relationship. An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the protocol and case report form (CRF) in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 30 minutes after each injection
Population: The SafAS population consisted of participants who had received study vaccine and for which safety data were scheduled to be collected.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 88 | 44
percentage of participants | 0 [0 to 4.1] | 0 [0 to 8.0]

2. Primary Outcome: Percentage of Participants With Solicited Injection-Site Reactions
Description: An AE was any untoward medical occurrence in a participant administered study vaccine and which did not necessarily have a causal relationship. A solicited reaction was an expected adverse reaction (AR) observed and reported under the conditions pre-listed in the protocol and CRF and included pain, erythema, and swelling. Injection site reaction was an AR at and around the injection site. Injection site reactions were commonly inflammatory reactions.
Time Frame: Up to 7 days after each injection
Population: The SafAS population consisted of participants who had received study vaccine and for which safety data were scheduled to be collected. Only those participants with data available were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 87 | 44
percentage of participants | 19.5 [11.8 to 29.4] | 29.5 [16.8 to 45.2]

3. Primary Outcome: Percentage of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" adverse reaction (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRF. Solicited systemic reactions included headache, fever, localized or topical manifestations that were not associated with the vaccination or administration site.
Time Frame: Up to 14 days after each injection
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 88 | 44
percentage of participants | 61.4 [50.4 to 71.6] | 72.7 [57.2 to 85.0]

4. Primary Outcome: Percentage of Participants With Unsolicited AE, Serious and Non-Serious AEs of Special Interest (AESIs)
Description: An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the protocol and CRF in terms of diagnosis and/or onset window post-vaccination. An AESI was one of scientific and medical concern specific to the study vaccine, for which ongoing monitoring, and rapid communication by the Investigator to the Sponsor was appropriate. The following were considered as serious AESI: serious hypersensitivity/allergic reactions occurring in all participants within 7 days after vaccination; serious viscerotropic disease occurring in all participants within 30 days after vaccination; serious neurotropic disease occurring in all participants within 30 days after vaccination; serious dengue disease requiring hospitalization occurring in all participants at any time during the study. The following were considered as non-serious AESIs, hypersensitivity/allergic reactions occurring in all participants within 7 days after vaccination.
Time Frame: Up to 28 days after each injection
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 88 | 44
percentage of participants
  Unsolicited AE | 55.7 [44.7 to 66.3] | 65.9 [50.1 to 79.5]
  Serious AESI | 0 [0 to 4.1] | 0 [0 to 8.0]
  Non-serious AESI | 4.5 [1.3 to 11.2] | 2.3 [0.1 to 12.0]

5. Primary Outcome: Percentage of Participants With Serious AEs (SAEs) and Hospitalized Virologically-Confirmed Dengue (VCD) Cases
Description: An AE was any untoward medical occurrence in a participant administered study vaccine and which does not necessarily have a causal relationship. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Hospitalized VCD cases were defined as an acute febrile illness with diagnosis of dengue requiring hospitalization. The confirmatory dengue diagnosis was performed through virological detection.
Time Frame: From the date of randomization until 6-month safety follow-up (approximately 38 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 88 | 44
percentage of participants
  SAE | 13.6 [7.2 to 22.6] | 15.9 [6.6 to 30.1]
  Hospitalized VCD Cases | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Geometric Mean Titers of Neutralizing Antibody Levels Against Each of the 4 Parental Dengue Virus Strains
Description: Dengue neutralizing antibody levels were measured by PRNT50. Serial, 2-fold dilutions of serum to be tested (previously heat-inactivated) were mixed with a constant challenge-dose of each dengue virus serotype 1, 2, 3 or 4. The presence of dengue virus infected cells was indicated by formation of plaques. A reduction in virus infectivity due to neutralization by antibody present in serum samples was detected. The reported value represented the highest dilution of serum at which >= 50% of dengue challenge virus (in plaque counts) was neutralized when compared to the mean viral plaque count in the negative control wells which represented the 100% virus load.
Time Frame: Baseline (Day 0) and 28 days after each injection
Population: The Full analysis set consisted of participants who received either CYD dengue vaccine or placebo and had blood sample drawn and valid post-injection serology results. Only data from the participants analyzed were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 87 | 44
Titer
  Serotype 1, Day 0: number analyzed (Participants) | 86 | 44
  Serotype 1, Day 0 | 176 [113 to 273] | 256 [142 to 464]
  Serotype 1, Day 28 | 589 [394 to 881] | 227 [131 to 393]
  Serotype 1, Day 211: number analyzed (Participants) | 84 | 44
  Serotype 1, Day 211 | 508 [350 to 736] | 260 [151 to 449]
  Serotype 1, Day 393: number analyzed (Participants) | 81 | 42
  Serotype 1, Day 393 | 535 [363 to 789] | 252 [142 to 447]
  Serotype 2, Day 0: number analyzed (Participants) | 86 | 44
  Serotype 2, Day 0 | 263 [177 to 390] | 426 [275 to 658]
  Serotype 2, Day 28 | 979 [750 to 1279] | 411 [288 to 586]
  Serotype 2, Day 211: number analyzed (Participants) | 84 | 44
  Serotype 2, Day 211 | 834 [639 to 1089] | 496 [331 to 741]
  Serotype 2, Day 393: number analyzed (Participants) | 81 | 42
  Serotype 2, Day 393 | 845 [623 to 1146] | 532 [368 to 771]
  Serotype 3, Day 0: number analyzed (Participants) | 86 | 44
  Serotype 3, Day 0 | 142 [98.2 to 205] | 233 [140 to 389]
  Serotype 3, Day 28 | 526 [390 to 709] | 202 [117 to 349]
  Serotype 3, Day 211: number analyzed (Participants) | 84 | 44
  Serotype 3, Day 211 | 383 [285 to 516] | 204 [123 to 336]
  Serotype 3, Day 393: number analyzed (Participants) | 81 | 42
  Serotype 3, Day 393 | 310 [237 to 404] | 179 [110 to 292]
  Serotype 4, Day 0: number analyzed (Participants) | 86 | 44
  Serotype 4, Day 0 | 67.4 [47.4 to 95.2] | 80.2 [49.5 to 130]
  Serotype 4, Day 28 | 489 [376 to 635] | 89.7 [58.3 to 138]
  Serotype 4, Day 211: number analyzed (Participants) | 84 | 44
  Serotype 4, Day 211 | 414 [321 to 535] | 109 [65.3 to 183]
  Serotype 4, Day 393: number analyzed (Participants) | 81 | 42
  Serotype 4, Day 393 | 354 [281 to 445] | 86.1 [54.0 to 137]

7. Secondary Outcome: Percentage of Participants With a Detected and Quantified CYD Dengue Vaccinal Viremia
Description: The percentage of participants with detected and quantified CYD dengue vaccinal viremia, i.e above the detection level as assessed by reverse transcription-polymerase chain reaction (RT-PCR) and for each of the 4 dengue serotypes after the first CYD dengue vaccine injection has been reported. Four RT-PCRs were used to perform quantitation and serotype identification of post-vaccinal serotype-specific dengue vaccine viremia from serum samples displaying a positive yellow fever (YF) RT-PCR result. The assay was performed only for YT RT-PCR-positive samples.
Time Frame: At 7 and 14 days post-injection 1
Population: The SafAS population consisted of participants who had received study vaccine and for which safety data were scheduled to be collected. Only data from the participants analyzed were reported.
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 12 | 0
percentage of participants
  Serotype 1, Detectable viremia, Day 7 | 8.3 |
  Serotype 1, Quantified viremia, Day 7 | 0 |
  Serotype 2, Detectable viremia, Day 7 | 0 |
  Serotype 2, Quantified viremia, Day 7 | 0 |
  Serotype 3, Detectable viremia, Day 7 | 0 |
  Serotype 3, Quantified viremia, Day 7 | 0 |
  Serotype 4, Detectable viremia, Day 7 | 41.7 |
  Serotype 4, Quantified viremia, Day 7 | 0 |
  Serotype 1, Detectable viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 1, Detectable viremia, Day 14 | 0 |
  Serotype 1, Quantified viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 1, Quantified viremia, Day 14 | 0 |
  Serotype 2, Detectable viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 2, Detectable viremia, Day 14 | 0 |
  Serotype 2, Quantified viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 2, Quantified viremia, Day 14 | 0 |
  Serotype 3, Detectable viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 3, Detectable viremia, Day 14 | 0 |
  Serotype 3, Quantified viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 3, Quantified viremia, Day 14 | 0 |
  Serotype 4, Detectable viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 4, Detectable viremia, Day 14 | 50.0 |
  Serotype 4, Quantified viremia, Day 14: number analyzed (Participants) | 2 | 0
  Serotype 4, Quantified viremia, Day 14 | 0 |

8. Secondary Outcome: Percentage of Participants With Clusters of Differentiation 4 (CD4) Count Decrease
Description: A decrease in CD4 count greater than 30 % assessed 28 days post-injection compared to the pre-injection value, not explained by non-adherence to antiretroviral therapy (ART) and not explained by any other possible etiology, and confirmed by a second test taken 4 weeks after the first (ie, approximately 2 months post-injection) showing the same value/trend.
Time Frame: From Day 28 to Day 393 (28 days after each injection)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 87 | 44
percentage of participants | 6.9 [2.6 to 14.4] | 2.3 [0.1 to 12.0]

9. Secondary Outcome: Percentage of Participants With Confirmed Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) Viral Load Increase
Description: A confirmed HIV viral load increase was defined as plasma HIV-1 RNA >1000 copies/milliliter (mL) 28 days post-injection after having been undetectable (< 50 copies/mL) pre-injection, not explained by non-adherence to ART and not explained by any other possible etiology and confirmed by a second test taken 4 weeks after the first (i.e, approximately 2 months post-injection) showing the same value/trend.
Time Frame: From Day 28 to Day 393 (28 days after each injection)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CYD Dengue Vaccine | Placebo
Number analyzed (Participants) | 88 | 44
percentage of participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of randomization until 6-month safety follow-up (approximately 38 months)
Description: Analysis was performed on SafAS population.
Arm/Group | CYD Dengue Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/88 | 0/44
Serious Adverse Events (participants affected / at risk) | 12/88 | 7/44
Other Adverse Events (participants affected / at risk) | 61/88 | 35/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine (N=88) | Placebo (N=44)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cd4 Lymphocytes Decreased (Investigations) | 10 (11) | 4 (5)
Viral Load Increased (Investigations) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine (N=88) | Placebo (N=44)
Asthenia (General disorders) | 27 (38) | 16 (18)
Injection Site Pain (General disorders) | 16 (22) | 13 (18)
Malaise (General disorders) | 32 (47) | 21 (27)
Covid-19 (Infections and infestations) | 6 (6) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 4 (4) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (39) | 18 (22)
Headache (Nervous system disorders) | 42 (67) | 28 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/28/NCT02741128/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT02741128/SAP_001.pdf